CLINICAL TRIAL: NCT01546870
Title: Coronary Artery Study in Pediatric Heart Transplantation
Acronym: CAS-POHT
Status: Withdrawn | Type: Observational
Why Stopped: never approved by IRB
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: ArkansasChRI
Record Dates: First submitted 2012-03-03; First posted 2012-03-07 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Transplant Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pediatric heart transplant recipients

SUMMARY:
Transplant coronary artery disease (TCAD) is a significant cause of morbidity and mortality in pediatric heart transplantation (PHT). Understanding the pathophysiology and early detection along with attempted medical management are crucial in preventing advancement of the disease and retransplantation or mortality. Coronary angiogram, although routinely used is insensitive to detect early TCAD. Measurement of fractional flow reserve (FFR), coronary flow reserve (CFR) and index of microvascular resistance (IMR) using a doppler pressure and flow intracoronary wire may be more sensitive in evaluating the integrity of coronary vasculature and thus detect pre clinical TCAD. To the best of the investigators knowledge, measurement of these parameters has not been previously reported in PHT.

ELIGIBILITY:
Inclusion Criteria:

* less than 21 years and above 7 years of age

Exclusion Criteria:

* clinically significant coronary artery disease on angiography and inability to undergo IVUS

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric heart transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Clinical coronary artery disease | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's hospital, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Fearon WF, Hirohata A, Nakamura M, Luikart H, Lee DP, Vagelos RH, Hunt SA, Valantine HA, Fitzgerald PJ, Yock PG, Yeung AC. Discordant changes in epicardial and microvascular coronary physiology after cardiac transplantation: Physiologic Investigation for Transplant Arteriopathy II (PITA II) study. J Heart Lung Transplant. 2006 Jul;25(7):765-71. doi: 10.1016/j.healun.2006.03.003. Epub 2006 May 24. PMID 16818118